CLINICAL TRIAL: NCT06404164
Title: Artificial Intelligence Pulmonary Watershed Terrain Navigation System for Lung Nodule Localization and Lung Function Preservation
Brief Title: Pulmonary Watershed Topographic Map Navigation for Lung Nodule Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Director, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Watershed
Record Dates: First submitted 2024-04-27; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Function Assessment; Disease Free Survival; NSCLC, Stage I
Keywords: Watershed Analysis; wedge resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Watershed analysis (Other)
  Interventions: Procedure: Wedge resection under watershed analysis method

INTERVENTIONS:
Procedure: Wedge resection under watershed analysis method — * Compare the preoperative 3D reconstruction model, and use electrocautery to directionally separate and expose the target artery;
    * Auxiliary devices (unlimited) to block the target artery, but should not be severed; ③ Peripheral intravenous injection of ICG, electrocautery to mark the border of counter-staining; ④ Evaluate the actual incisal margin according to the preoperative planning, and use the cutting stapler to wedge resection of the pulmonary nodule

SUMMARY:
A method of ICG counterstaining localization under target artery occlusion without cutting，It's a new method of localization of small pulmonary nodules.

DETAILED DESCRIPTION:
1. This technology can replace part of CT puncture-guided positioning, which not only saves CT positioning costs for patients, but also saves time and space resources in CT room;
2. The target artery occlusion technique does not cut off the blood vessels, and the operation is still a wedge resection. Compared with the standard segmentectomy/subsegmentectomy, the steps of cutting off the veins and bronchial tubes are reduced, the operation time is shortened, and the turnover rate is improved.
3. There is less damage to the lung tissue, and the lung function is well preserved. The patients can be discharged in an average of 3 days after the operation, which improves the bed turnover efficiency of the department.

ELIGIBILITY:
Inclusion Criteria:

1. <1cm CTR≤0.75; <1.5cm CTR≤0.5; <2cm CTR≤0.25 Lung nodules
2. The tumor center is located in the peripheral 2/3 area of the lung field
3. Preoperative analysis and planning of watershed by 3D reconstruction
4. Clinically assessed as cT1aN0M0 stage IA1/cT1bN0M0 stage IA2 (eighth edition), clinically resectable

Exclusion Criteria:

1. No surgical video, no postoperative gross specimen and related distance measurement records
2. The incision edge does not exceed the target nodule diameter from the nodule edge
3. The resection range exceeds 50% of the preoperative planning
4. Postoperative pathological staging non-pT1aN0M0 IA1 stage/pT1bN0M0 IA2 stage (eighth edition)
5. Any situation where the investigator feels the need for extended resection
6. Patients with chronic diseases (such as COPD, pulmonary fibrosis, silicosis) that can cause loss of lung function in patients at risk of progression or potential progression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Lung fuction | 1month 3month 1year
  testing FEV1 and FVC with MIR Spirolab

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No